CLINICAL TRIAL: NCT06181474
Title: Assessment of the Symptomatic Burden of Patients With Advanced Chronic Liver Disease. Correlation Between the Model for End-Stage Liver Disease (MELD)-Na and the Edmonton Symptom Assessment System Scale (ESAS).
Brief Title: MELD ESAS Evolution: Assessment of the Symptomatic Burden of Patients With Advanced Chronic Liver Disease
Acronym: MELDESAS
Status: Completed | Type: Observational
Sponsor: Unidade Local de Saúde de Matosinhos, EPE (Other)
Responsible Party: Principal Investigator, Hugo Miguel Oliveira, Principal Investigator, Universidade do Porto
Other Study IDs: ULSM_131/CES/JAS
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-03

CONDITIONS: Palliative Care; End Stage Liver DIsease
Keywords: Hepatology; End Stage Liver Disease; Palliative Care
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: ESAS — Observation of symptoms

SUMMARY:
The goal of this observational study is to understand if there is a correlation between the evolution of MELD-Na and symptomatic burden of patients with advanced chronic liver disease.

All patients with chronic liver disease will be invited to participate in the study. Patients will be followed prospectively with assessment of their MELD-Na score and symptom burden, according to the Edmonton Symptom Assessment System scale.

DETAILED DESCRIPTION:
1. Methodology - Prospective observational study
2. Population - All patients with chronic liver disease followed in the Matosinhos Local Health Unit after their first episode of decompensation or are diagnosed with hepatocellular carcinoma in stage C or D of the Barcelona Liver Clinic Cancer will be invited to participate in the study.

   All patients who do not sign consent to participate, patients under 18 years of age and patients who present a recurrent degree of encephalopathy, according to the West-Haven scale, equal or greater than 2, will be excluded.
3. Sample - Non-probabilistic for convenience
4. Data collection instrument - Patients will be followed prospectively with quarterly assessment, or after each episode of decompensation, of their MELD-Na score and symptom burden, according to the Edmonton Symptom Assessment System scale (ESAS), with introduction of 3 other symptoms prevalent in patients with chronic liver disease: sexual dysfunction sexual, cramps and pruritus. The minimum analysis for each patient will be 2 assessments.

   All symptoms greater than 5 points will be considered moderate to severe and formal referral to the palliative care team will be discussed with the patient and their attending physician. Subsequently evaluating its effectiveness in symptomatic control.
5. Aims - This observational study will try to understand if there is a correlation between the evolution of MELD-Na and symptomatic burden of patients with advanced chronic liver disease. As well as the influence that the implementation of palliative care have on symptom burden of advanced chronic liver disease patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic liver disease

Exclusion Criteria:

* do not sign consent to participate
* patients under 18 years of age
* patients who present a recurrent degree of encephalopathy, according to the West-Haven scale, equal or greater than 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic liver disease followed in the Matosinhos Local Health Unit after their first episode of decompensation or are diagnosed with hepatocellular carcinoma in stage C or D of the Barcelona Liver Clinic Cancer will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
MELD ESAS | 1 year
  Evaluate and correlate the evolution of MELD-Na and ESAS on advanced chronic liver disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Hugo Miguel Oliveira, Matosinhos Municipality, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira HM, Ribeiro F, Lopes G, Frias E, Andrade F, Guiomar V, Eiras E, Rego F, Nunes R. Symptom burden in end-stage liver disease: a prospective cohort study of the symptoms experienced by patients and the role of palliative care. Therap Adv Gastroenterol. 2025 Jul 13;18:17562848251353624. doi: 10.1177/17562848251353624. eCollection 2025. PMID 40661221